CLINICAL TRIAL: NCT03568448
Title: Monitoring Response to Neoadjuvant Chemotherapy (NAC) in HER2 Negative Breast Cancer (HNBC) Using High-speed MR Spectroscopic Imaging (MRSI)
Brief Title: Monitoring Response to Neoadjuvant Chemotherapy in HER2 Negative Breast Cancer Using High-speed MR Spectroscopic Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 1607
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: HER2 Negative Breast Cancer
Keywords: HER2 negative breast cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Response monitoring (no intervention) — Response monitoring (no intervention)

SUMMARY:
The study will assess whether changes in total choline concentration [tCho] during neoadjuvant chemotherapy (NAC) are predictive of pathologic complete response (pCR) in patients with HER2 negative breast cancer (HNBC) appropriate for NAC, and compare these findings with dynamic contrast enhanced magnetic resonance imaging (DCE-MRI). The objective is to assess the predictive value of changes in the concentration and spatial extent of tCho within the tumor during NAC.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the correlation of serial high-speed MRSI of [tCho] with pCR following NAC in women with HNBC. The endpoint is the pCR.

Hypothesis 1: Changes in [tCho] early during NAC (from 24 hours after the start of the first cycle until the start of the 2nd cycle of NAC) are predictive of pathologic response (using quantitative metrics of Residual Cancer Burden (RCB)1 and/or CPS+EG score 2 and radiologic response (change in lesion size on DCE-MRI).

Hypothesis 2: Decreases in [tCho] within the tumor precede decreases in tumor volume on DCE-MRI, thus enabling earlier discrimination between responders from non-responders. The primary objective of the study is to assess the correlation of serial high-speed magnetic resonance spectroscopic imaging (MRSI) of [tCho] with pCR following NAC for HNBC. The secondary objective is to compare the time course of [tCho] on serial high-speed MRSI and tumor volume on serial DCE-MRI for predicting early NAC treatment response in HNBC.

Subjects' participation will start approximately 2 weeks before initiation of neoadjuvant therapy and end after surgery.

Patients will undergo up to 5 MRI scans in total as 2 are clinical MRIs and 3 are research scans. The clinical pretreatment MRI scan and a post treatment MRI scan are standard and will be ordered at the discretion of the treating provider.The post treatment MRI is done after clinical response and before surgery. This helps guide the surgeon about what amount of tissue should be removed at surgery. The minimum time between clinical and research MRI scans is 24 hours.

The 3 research MRIs will be performed on a 3T Siemens scanner equipped with 16 channel Hologic breast coil. Breast anatomy will be imaged using a bilateral localizer, an axial T 2-weighted turbo-spin-echo scan, and a fat-suppressed T1-weighted sagittal gradient echo scan. Dynamic non-fat-suppressed T1-weighted axial 3D GRE scans are collected before and with 20s delay at four time points after Gd-HP-DO3A administration (total scan time: 7.5 min). Subtraction images are created using the pre-contrast image as the mask. A diffusion weighted multi-slice EPI scan will be performed to compute apparent diffusion coefficient (ADC) maps online (total scan time: 3:14 min). An axial low-resolution multi-slice multi-echo gradient echo scan will be performed to compute field maps for slice and laterality specific auto-shimming. Spectroscopic imaging will be performed using 3D PEPSI.

The MR measurement protocol will be performed at 3 time points: (1) prior to treatment typically several days before NAC (ideally 24h before NAC) (MRSI, DW-MRI, DCE-MRI), (2) 20-52 hours after the beginning of the first cycle of NAC (MRSI, DW-MRI), and (3) between the first and second cycle of NAC (MRSI, DW-MRI, DCE-MRI).

Surgery will be performed within 3 to 12 weeks of last chemotherapy. RCB will be obtained from the final pathologic findings.

ELIGIBILITY:
Inclusion Criteria:

* Have a biopsy proven HER2 negative (by IHC or FISH) breast cancer per standard clinical criteria (per ASCO-CAP guidelines). Although patients with hormone-receptor positive (ER+ and/or PR+) disease will be included, patients with tumor features indicative of luminal A intrinsic sub-type will be excluded from this study. Excluding features are:

  * Patients with Grade 1 breast cancers, as assessed by local standard criteria, will be excluded from participation.
  * Patients with strongly ER AND PR positive breast cancer, defined as >75% positive staging for BOTH markers by IHC, will be excluded from participation.
* Stage of disease that is appropriate for standard NAC (any combination of T2 to T4, N0 to N3 that would comprise stage IIA to IIIB disease). Patients with inflammatory carcinoma or stage IIIC disease who are deemed inoperable at the outset, but appropriate for NAC are excluded in this study since there is no guarantee they can be converted to operability following NAC; thus precluding assessment of pCR.
* Medically fit for NAC as per good clinical practice and per the treating physician's judgment.
* Age > or = to 18 years AND able to provide informed consent.
* Women of childbearing potential must be willing and able to use effective means of contraception. A female of childbearing potential is any woman who has not undergone a hysterectomy or bilateral oophorectomy or has not had menses at any time in the preceding 12 consecutive months.
* Able to undergo standard clinical MRI exams PLUS additional 30 minutes longer (total scan time is 50 to 60 minutes).

Exclusion Criteria:

* Pregnant or lactating women.
* Body contains foreign items posing an issue of MRI safety, such as intra-ocular metallic foreign bodies, MRI incompatible devices such as pacemakers and cochlear implants, and other MRI incompatible devices.
* Obesity (Body Mass Index [BMI] > 40) or inability to fit into the standard MRI gantry.
* Suffer from back pain, claustrophobia, seizures, panic disorder and/or other medical disorders severe enough that would prevent them from completing a standard clinical MRI study (30 min) + 30 mins for the research scans. If applicable, patients may take a mild anxiolytic (e.g., lorazepam) if deemed appropriate by their treating physician.
* Patients with stage IV disease (gross metastasis or documented M1 disease) and stage of disease excluded above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible female breast cancer patients receiving treatment at the University of New Mexico Comprehensive Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the correlation of serial high-speed MRSI of [tCho] with pCR following NAC | Patient will begin participation 2 weeks prior to initiation of NAC and will complete participation at the time of surgery, estimated to be 4-6 months total participation duration.
  In this study changes in total choline concentration [tCho] during neoadjuvant chemotherapy (NAC) will be evaluated by performing a high-speed magnetic resonance spectroscopic imaging (MRSI) at baseline prior to first cycle NAC, after first cycle NAC, and prior to second cycle NAC.

SECONDARY OUTCOMES:
Assess the correlation of serial high-speed MRSI of [tCho] with response to NAC | Patient will begin participation 2 weeks prior to initiation of NAC and will complete participation at the time of surgery, estimated to be 4-6 months total participation duration.
  The endpoint is response as assessed by the validated quantitative metrics of Residual Cancer Burden (RCB) and/or CPS+EG score.
Compare the time course of [tCho] on serial high-speed MRSI and tumor volume on serial DCE-MRI for predicting early NAC treatment response | Patient will begin participation 2 weeks prior to initiation of NAC and will complete participation at the time of surgery, estimated to be 4-6 months total participation duration.
  Outcome measured will be total choline concentration [tCho] as assessed via serial high-speed magnetic resonance spectroscopic imaging (MRSI) .

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Posse, PhD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No